CLINICAL TRIAL: NCT06392529
Title: Efficacy of Voriconazole Loaded Spanlastics Gel Versus Clotriamazole Cream on Treating Vulvovaginal Candidasis
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Raghda R.S. Hussein, Assistant Professor of Clinical Pharmacy and Head of Department, Beni-Suef University
Other Study IDs: REC-H-PhBSU-24009
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Voriconazole Group
  Interventions: Drug: Voriconazole Powder
- Clotriamazole group
  Interventions: Drug: Voriconazole Powder

INTERVENTIONS:
Drug: Voriconazole Powder — The drug will be topically applied for vagina of patients suffering from vaginal Candidasis albican

SUMMARY:
To investigate and compare the efficacy of voriconazole loaded spanlastics (VCZ loaded SPs) optimum gel formula (F2 VCZ loaded SP gel) versus Clotrimazole cream in treating candida albicans causing vulvovaginal candidiasis for different durations of 3 days and 5 days.

DETAILED DESCRIPTION:
The current study will be prospective controlled randomized clinical trial. 28 female patients suffering from vulvovaginal candidiasis will be enrolled in the following 2 groups:

Gp 1 (Test group): including 14 patients with vulvovaginal candidiasis albicans that will be randomized in the following subgroups:

Gp 1a: will be treated with F2 VCZ loaded SP gel for 3 days. Gp 1 b: Will be treated with F2 VCZ loaded SP gel for 5 days. Gp 2 (Control group): including 14 patients with vulvovaginal candidiasis albicans will be randomized in the following sub groups Gp 2 a: will be treated with the Clotrimazole cream available in the market for 3 days.

Gp 2 b: Will be treated with the Clotrimazole cream available in the market for 5 days.

Smears will be taken from the patients before starting the therapeutic protocol and after finishing it. Compliance of the patients to the creams will be assesses

ELIGIBILITY:
Inclusion Criteria:

* Female patients aging from 20 t0 40 years old suffering from vulvovaginal candidiasis caused by albicans species.

Exclusion Criteria:

* Pregnant women, female suffering from vulvovaginal candidiasis caused by other species rather than C. albicans.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Female patients suffering from vulvovaginal candidiasis albicans
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
efficacy of nano voriconazole versus Clotrimazole in Treatment of vaginal candidiasis albicans and removal of symptoms | 1Month
  To assess and compare the efficacy of nano voriconazole versus Clotrimazole in Treatment of vaginal candidiasis albicans in 3 and 5 days via smear cultures

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University Teaching Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided